CLINICAL TRIAL: NCT05910918
Title: Effect of Intensive Care Nurses' Training Package on the Safety Culture of Critically Ill Geriatric Patients:Findings and Implications for Clinical Practice
Brief Title: Intensive Care Nurses' Training Package on the Safety Culture of Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, assistant professor, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1522102022
Record Dates: First submitted 2023-02-19; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Safety
Keywords: Geriatric Patients; Critically ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Care Nurses' Training Package (Experimental): For the study group, the researcher will explain the method of the training package program application to critical care nurses as follows; firstly, the researchers will assess the nurses' roster, then the researchers will classify the subjects into groups in order to conduct the training package for a group of them while the other subjects taking care of the patients in the intensive care units and repeat the same session to the others in the same manner.
  Interventions: Behavioral: Intensive Care Nurses' Training Package
- comparison group (Active Comparator): for the comparison group receive the general intensive care rules manual for routine care.
  Interventions: Behavioral: Intensive Care Nurses' Training Package

INTERVENTIONS:
Behavioral: Intensive Care Nurses' Training Package — For the study group, the researcher will explain the method of the training package program application to critical care nurses as follows; firstly, the researchers will assess the nurses' roster, then the researchers will classify the subjects into groups in order to conduct the training package for a group of them while the other subjects taking care of the patients in the intensive care units and repeat the same session to the others in the same manner.

SUMMARY:
This study aims to determine the effect of intensive care nurses' training package on the safety culture of critically ill geriatric patients.

Study hypothesis:

Intensive care nurses who receive the proposed training package exhibit higher scores on critically ill geriatric patients' safety culture awareness than those who do not receive it.

DETAILED DESCRIPTION:
The researchers will prepare the proposed nurses' training package program. The program will be planned to be carried out in 10 sessions that will be classified into; sessions regarding knowledge about the age-related changes affecting elderly patients that should be considered while caring for them and how to care for and maintain the safety of the critically ill geriatric patients. The researchers will prepare an illustrative PowerPoint presentation of each study program's session.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 years and above.
* provide direct care for critically ill geriatric patients.
* work for at least 1 month in the unit.

Exclusion Criteria:

• not involved in patient care.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Intensive Care Nurses' Awareness of the Critically Ill Geriatric Patients' Safety Culture Questionnaire | 2 weeks
  This tool will assess the intensive care nurses' awareness of critically ill geriatric patients' safety culture. It will include items that will be categorized into four subscales namely, intensive care nurses' knowledge, attitude, and practices of caring for critically ill geriatric patients and the critical care unit work environment. The nurses have to respond to the items using a 3-point Likert scale. The total score of the items will be summed and higher scores will indicate greater nurses' awareness of critically ill geriatric patients' safety culture.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, Study Chair — Egypt Faculty of Nursing Alexandria, Egypt
Locations (2):
- Egypt (2):
  - Rasha Eweida, Alexandria
  - Faculty of Nursing, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen YL, Angus DC, Boumendil A, Guidet B. The challenge of admitting the very elderly to intensive care. Ann Intensive Care. 2011 Aug 1;1(1):29. doi: 10.1186/2110-5820-1-29. PMID 21906383
- [Background] Laake JH, Dybwik K, Flaatten HK, Fonneland IL, Kvale R, Strand K. Impact of the post-World War II generation on intensive care needs in Norway. Acta Anaesthesiol Scand. 2010 Apr;54(4):479-84. doi: 10.1111/j.1399-6576.2009.02170.x. Epub 2009 Nov 23. PMID 19930244
- [Background] Bagshaw SM, Webb SA, Delaney A, George C, Pilcher D, Hart GK, Bellomo R. Very old patients admitted to intensive care in Australia and New Zealand: a multi-centre cohort analysis. Crit Care. 2009;13(2):R45. doi: 10.1186/cc7768. Epub 2009 Apr 1. PMID 19335921
- [Background] Boumendil A, Somme D, Garrouste-Orgeas M, Guidet B. Should elderly patients be admitted to the intensive care unit? Intensive Care Med. 2007 Jul;33(7):1252. doi: 10.1007/s00134-007-0621-3. Epub 2007 Apr 3. PMID 17404703